CLINICAL TRIAL: NCT04638517
Title: The TELO-SCOPE Study: Attenuating Telomere Attrition With Danazol. Is There Scope to Dramatically Improve Health Outcomes for Adults and Children With Pulmonary Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data Safety Monitoring Board recommended cessation due to futility
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TELO-SCOPE
Record Dates: First submitted 2020-11-04; First posted 2020-11-20 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Fibrosis; Telomere Shortening; Telomere Disease; Dyskeratosis Congenita
MeSH Terms: conditions — Pulmonary Fibrosis; Dyskeratosis Congenita | interventions — Danazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Danazol (Active Comparator): 800mg daily in two divided doses orally for 12 months. In subjects who have difficulty tolerating danazol / placebo, the dose will be reduced by 200mg/day and side effects will be reassessed. If symptoms related to the study drug persist, subsequent 200mg/day dose reductions will be allowed until a tolerated dose is achieved. Background antifibrotic therapy is allowed.
  Interventions: Drug: Danazol
- Placebo (Placebo Comparator): Matching placebo capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Danazol — Danazol up to 800mg daily in two-divided doses.
  Arms: Danazol
Drug: Placebo — Matching placebo.
  Arms: Placebo

SUMMARY:
TELO-SCOPE is a national, multi-centre, double-blind, placebo-controlled, randomised (2:1) trial which will test the hypothesis that, compared to placebo, the addition of danazol to standard of care in pulmonary fibrosis associated with short telomeres is safe and will result in reduced telomere attrition.

DETAILED DESCRIPTION:
TELO-SCOPE is a national, multi-centre, double-blind, placebo-controlled, randomised trial which will be conducted in subjects aged >5 years with a multi-disciplinary diagnosis of pulmonary fibrosis and with age-adjusted telomere length below the 10th centile in adults; and for children (age < 16 years), a confirmed diagnosis of Dyskeratosis Congenita (DC). Consenting participants who meet all other inclusions and no exclusions will be randomised (n=50, 2:1 (danazol:placebo)) to receive danazol (maximum tolerated dose (up to 800mg daily, two-divided doses) or matched placebo, for 12 months in addition to standard of care background therapy. The primary outcome is change in telomere length at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged >5 years, able to take capsules orally.
2. Fibrosing interstitial pneumonia (Idiopathic PF, idiopathic non-specific interstitial pneumonia, chronic hypersensitivity pneumonitis, pleuroparenchymal fibroelastosis, unclassifiable interstitial lung disease (ILD)) diagnosed according to the current international guidelines.
3. Age-adjusted peripheral blood leukocyte telomere length < 10th centile on Flow-FISH.
4. FVC > 40% predicted.
5. DLCO > 25% predicted.
6. If receiving background pirfenidone / nintedanib, stable dose for 28 days prior to screening.
7. Able to understand and sign a written informed consent form (or legally authorised representative).
8. Agreement to use a medically approved form of non-hormonal contraception (if of child-bearing potential) (noting that oral contraceptives are advised not to be used concurrently with danazol).

Exclusion Criteria:

1. Actively or imminently listed for lung transplantation.
2. Undergone, awaiting, or likely to require bone marrow transplantation within 12 months.
3. Concurrent enrolment in another study.
4. Females with a positive pregnancy test at screening or currently breastfeeding.
5. Pelvic infection.
6. Past jaundice with oral contraceptives.
7. Undiagnosed abnormal genital bleeding.
8. Undiagnosed ovarian/uterine masses
9. Any history of malignancy likely to result in significant disability or likely to require significant medical or surgical intervention within the next 12 months.
10. History of androgen-dependent tumour.
11. Any condition other than PF that, in the opinion of the investigator, is likely to result in the death of the participant within the next 12 months.
12. History of end-stage liver disease or ALT or AST > 3 times the upper limit of normal.
13. History of end-stage kidney disease requiring dialysis.
14. Markedly impaired cardiac function.
15. Known increased risk of or history of thromboembolism (e.g. Factor V Leiden, Protein C or S deficiency).
16. Uncontrolled hypertension.
17. Uncontrolled lipoprotein disorder.
18. Poorly-controlled diabetes mellitus.
19. History of marked or persistent androgenic reaction to previous gonadal steroid therapy.
20. History of epilepsy induced or worsened by previous gonadal steroid therapy.
21. History of raised intracranial pressure.
22. Known intolerance to danazol.
23. Porphyria.
24. Use of any of the following agents within 28 days before screening: danazol or other androgen therapy, warfarin or other anticoagulant, carbamazepine, phenytoin, investigational therapy, cytotoxic therapy, tacrolimus, cyclosporine.
25. Professional singer due to potential for voice change.
26. Competitive athletes.
27. Prostate specific antigen (PSA) above the upper limit of normal (adult males only).

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Change in absolute telomere length from baseline (base pairs) | 12 months
  Telomere length will be measured in absolute terms (base pairs) using the telomere shortest length assay (TeSLA).

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events | 12 months
Number of Participants With Death or Non-Elective Hospitalisation | 12 months
Change in telomere length from baseline to 3, 6 and 9 months (base pairs) | 3, 6 and 9 months
Change in forced vital capacity (FVC) at 6 and 12 months | 6 and 12 months
  FVC is measured as the volume of air exhaled during spirometry.
Change in diffusing capacity for carbon monoxide at 6 and 12 months | 6 and 12 months
  DLCO is a measurement of the of the lung's gas transfer ability.
Change in 6-minute walk distance from baseline | 12 months
Change in Leicester cough questionnaire (LCQ) from baseline | 12 months
Change in King's Brief Interstitial Lung Disease Questionnaire (K-BILD) from baseline | 12 months
Change in Parent cough-specific quality of life (PCSQoL) from baseline | 12 months

CONTACTS AND LOCATIONS:
Locations (9):
- Australia (9):
  - John Hunter Hospital, Newcastle, New South Wales
  - Sydney Children's Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - The Children's Hospital Westmead, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred, Melbourne, Victoria
  - The Austin, Melbourne, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be analysed and shared with collaborators with the plan to publish the results.

REFERENCES:
- [Derived] Mackintosh JA, Pietsch M, Lutzky V, Enever D, Bancroft S, Apte SH, Tan M, Yerkovich ST, Dickinson JL, Pickett HA, Selvadurai H, Grainge C, Goh NS, Hopkins P, Glaspole I, Reynolds PN, Wrobel J, Jaffe A, Corte TJ, Chambers DC. TELO-SCOPE study: a randomised, double-blind, placebo-controlled, phase 2 trial of danazol for short telomere related pulmonary fibrosis. BMJ Open Respir Res. 2021 Dec;8(1):e001127. doi: 10.1136/bmjresp-2021-001127. PMID 34857525